CLINICAL TRIAL: NCT02380586
Title: A National Survey on Obstetric Anesthesia and Analgesia Care - International
Brief Title: Obstetric Anaesthesia And Analgesia Month Attributes - International
Acronym: OBAAMA-INT
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Charles University, Czech Republic (Other); Masaryk University (Other); General University Hospital, Prague (Other); Czech society of anesthesiology, resuscitation a intensive care - ČLS JEP (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, MD, Ph.D, Brno University Hospital
Other Study IDs: MU_IBA1026
Record Dates: First submitted 2015-02-28; First posted 2015-03-05 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Obstetric Anesthesia Care
MeSH Terms: interventions — Anesthesia, Obstetrical; Analgesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women in labor undergoing anesthesia care: Women in labor undergoing anesthesia care
  Interventions: Procedure: Obstetric anesthesia and analgesia

INTERVENTIONS:
Procedure: Obstetric anesthesia and analgesia — All anesthesia procedures during labor: labor analgesia, anesthesia for Cesarean section, anesthesia for procedures in third stage of labor

SUMMARY:
A national survey of current practices, preferred drug and technique choices for obstetric anesthesia and analgesia in Czech Republic and Slovak Republic.

DETAILED DESCRIPTION:
A one month-long project monitoring an obstetric anesthesia practices in obstetric/anesthesia departments throughout the Czech Republic.

Electronic Case Report Form (eCRF) is used to collect data on all obstetric anesthesia procedures in peripartal period and obstetric and anesthesia complications. All consecutive cases in each participating center during the study period are recorded. Each record is related to parturient and contains the following sections: history, form of labour analgesia, type of anesthesia for Cesarean section and anesthesia in third stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Women in labor undergoing anesthesia care

Exclusion Criteria:

* not meeting inclusion criteria

Ages: 16 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women in labor
Sampling Method: Non-Probability Sample
Enrollment: 3040 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
A national survey of current practice of obstetric anesthesia and analgesia in Czech Republic and Slovak Republic | Parturition period, up to 24 hours after labor
  Monitoring of all obstetric anesthesia procedures in peripartal period and anesthesia complications: history, form of labour analgesia, type of anesthesia for Cesarean section and anesthesia in third stage of labor.

SECONDARY OUTCOMES:
Types of anesthesia a analgesia in peripartal period | Parturition period, up to 24 hours after labor
  To describe current practice a complications related to peripartal anesthesia care

OTHER OUTCOMES:
Complications related to obstetric anesthesia care | Parturition period, up to 24 hours after labor
  To describe current practice a complications related to peripartal anesthesia care

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, MD, Ph.D, Study Chair — FN Brno
Locations (1):
- Faculty Hospital Brno, Brno, Czech Republic, Czechia

REFERENCES:
- [Derived] Harazim H, Stourac P, Blaha J, Grochova M, Klozova R, Noskova P, Seidlova D, Richterova S, Svoboda M, Jarkovsky J, Silova X, Jezova B, Steinbach J, Zemanek M, Mannova J, Slavik J, Novakova Z, Misakova L, Firment J. The influence of mode of anaesthesia for caesarean delivery on neonatal Apgar scores in the Czech Republic and Slovakia: secondary analysis of the results of an international survey in 2015. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2019 Jun;163(2):147-154. doi: 10.5507/bp.2019.008. Epub 2019 Apr 9. PMID 30976125